CLINICAL TRIAL: NCT05170256
Title: HERES Trial: Trastuzumab and Standard Treatment With Chemo- and Immunotherapy as First Line Treatment for HER2 Positive Esophageal Squamous Cell Carcinoma Patients
Brief Title: Trastuzumab and Standard Treatment With Chemo- and Immunotherapy as First Line Treatment for HER2 Positive Esophageal Squamous Cell Carcinoma Patients
Acronym: HERES
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Morten Mau-Sørensen (Other)
Collaborators: Odense University Hospital (Other); Aalborg University Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Morten Mau-Sørensen, MD PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-003415-26
Record Dates: First submitted 2021-11-24; First posted 2021-12-27 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Esophageal Squamous Cell Carcinoma; HER-2 Protein Overexpression; HER-2 Gene Amplification
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Trastuzumab

STUDY DESIGN:
Intervention Model Description: The study is a two-staged single arm national phase II trial
  * Stage 1: 17 patients
  * Stage 2: 7 patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — Addition of trastuzumab to standard treatment (fluoropyrimidine/platinum doublet with pembrolizumab)

SUMMARY:
The study aims to determine the efficacy of trastuzumab added to standard treatment (fluoropyrimidine/platinum doublet with pembrolizumab) in patients with HER2 positive Esophageal squamous cell carcinoma (ESCC) determined by 6 months progression free survival (PFS) (RECIST 1.1).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age ≥18 years
3. Inoperable locally advanced or metastatic squamous cell carcinoma of the esophagus not amenable for curative intended therapy
4. HER2 positive defined as IHC2+ and FISH amplification ratio ≥2 or IHC3+
5. ECOG PS <2
6. Baseline left ventricular ejection fraction > 50% measured by echocardiography or MUGA
7. Adequate bone marrow function and organ function:

   1. Hematopoietic function:
   2. Leucocytes > 3.0 x 109/l, neutrocytes > 1.5 x 109/l and thrombocytes > 100 x 109/l
   3. Serum bilirubin < 1.5 × upper limit of normal (ULN); and AST/ALT < 2.5 × ULN (or < 5 × ULN in patients with liver metastases).
8. Creatinine clearance > 30 ml/min

Exclusion Criteria:

1. Prior systemic treatment with non-curative intent including HER2-targeting drugs. Prior neoadjuvant and adjuvant therapies as well as palliative radiotherapy are allowed
2. Significant medical illness that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate study treatment
3. Congestive heart failure (New York Heart Association (NYHA) class 3+4); uncontrolled angina pectoris; poorly controlled hypertension (systolic BP > 180 mmHg or diastolic BP > 100 mmHg); or high-risk uncontrollable arrhythmias.
4. Patients with severe dyspnoea at rest due to complications of advanced malignancy or requiring supplementary oxygen therapy.
5. Patients with known hypersensitivity to trastuzumab or any of the study drugs, murine proteins, or to any of the excipients
6. Symptomatic brain metastases uncontrolled by corticosteroids or carcinomatous meningitis
7. Homozygosity or compound heterozygosity for more than one gene variant of dihydropyrimidine dehydrogenase (DPD) known to cause major reduced metabolism of 5-FU derivates OR plasma uracil > 150 ng/ml are not eligible. Patients with minor DPD insufficiency are allowed provided that local guidelines for administration of 5-FU are followed.
8. Any other cancer (excluding low risk prostate cancer, carcinoma in situ and radically operated localised squamous skin cancer) with clinical activity within the last 2 years
9. Other current cancer treatments except for anti-hormone and anti-resorptive treatment of bone metastasis.
10. Allopurinol, phenytoin, warfarin treatment is not allowed. Non vitamin K oral anticoagulants (NOAK) and low molecular weight (LMW) heparin is allowed
11. Pregnancy or breast-feeding
12. Positive serum pregnancy test in women of childbearing potential.
13. Subjects with reproductive potential not willing to use an effective method of contraception under and 3 months after participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) . | 6 months
  PFS according to RECIST 1.1

SECONDARY OUTCOMES:
Response rate according to RECIST 1.1 | Best response during 6 months follow-up
  Partial, complete and overall response rate according to RECIST 1.1
Frequency of AEs assessed by NCI CTCAE, v. 5.0 | During minimum 6 months follow-up
  Safety and tolerability of trastuzumab, pembrolizumab and a fluoropyrimidine/platinum assessed by NCI CTCAE, v. 5.0
Overall survival | 6 months
  Time to death of all causes

OTHER OUTCOMES:
Change in amplified HER2 in ctDNA during treatment | During mininum 6 months follow-up
  Clinical utility of measurements of amplified HER2 in ctDNA as a monitoring tool of treatment with 5-FU platinum, trastuzumab and pembrolizumab
Frequency of germeline Fc Gamma Receptor polymorphisms | During minimum 6 months follow-up
  Predictive value of Fc Gamma Receptor polymorphisms in ESCC patients receiving
Frequency of PD-L1 status by CPS score | During minimum 6 months follow-up
  PD-L1 status by CPS score

CONTACTS AND LOCATIONS:
Overall Officials: Lene Baeksgaard, MD PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Dept of Oncology, Rigshospitalet, Copenhagen, Region H
  - Onkologisk Afdeling R, Odense University Hospital, Odense, Region Syd

IPD SHARING:
Plan to Share IPD: Undecided